CLINICAL TRIAL: NCT04567901
Title: Using the Geriatric Nutritional Risk Index (GNRI) to Evaluate the Influence of Nutrition on the Mortality of Trauma Patients
Brief Title: GNRI and Influence of Nutrition on the Mortality of Trauma Patients
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202001446B0
Record Dates: First submitted 2020-09-21; First posted 2020-09-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Trauma Injury
MeSH Terms: conditions — Accidental Injuries | interventions — Death Domain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trauma Patients: The enrolled patients experienced trauma from different injuries and were hospitalized for treatment and admitted to the ICU. 700 older trauma patients (age equal to or more than 65 years) were finally included in the study.
  Interventions: Other: Death; Other: Survive

INTERVENTIONS:
Other: Death — Mortality group
Other: Survive — Survival group

SUMMARY:
The geriatric nutritional risk index (GNRI) is a simple and efficient tool to assess the nutritional status of patients with malignancies or after surgery. Because trauma patients constitute a specific population that generally acquires accidental and acute injury, this study aimed to identify the association between the GNRI at admission and mortality outcomes of older trauma patients in the intensive care unit (ICU).

DETAILED DESCRIPTION:
The nutritional risk index (NRI) is a screening method that was primarily developed to identify older patients with malnutrition. It consists of serum albumin levels as well as body weight measurements. However, even under professional care, the usual body weight is often not documented for older patients. To determine the usual body weight of older patients, the geriatric nutritional risk index (GNRI) was introduced in 2005 by Bouillanne et al - the formula included a combination of serum albumin levels and the ratio of body weight to ideal body weight. The GNRI formula replaces the usual body weight in the NRI formula with the ideal body weight, calculated using the Lorentz formula. Although the GNRI was developed using the data of patients who were admitted to a geriatric rehabilitation care unit, it was found to be a strong prognostic factor for certain malignancies and a simple, objective, and quick method to determine the nutritional status of patients and long-term postoperative outcomes and the correlation between these elements. Using this simple calculation, it is possible to evaluate the nutritional status of critically ill patients with acute respiratory distress syndrome in the intensive care unit (ICU). Considering that trauma patients constitute a specific population, as injuries generally occur accidentally and acutely, it is important to determine whether the GNRI can be used to link nutritional status and outcomes in trauma patients. Therefore, this study aimed to identify the association between GNRI at admission and mortality outcomes of older trauma patients in the ICU.

ELIGIBILITY:
Inclusion Criteria:

* trauma from different injuries
* hospitalized for treatment
* admitted to the ICU

Exclusion Criteria:

* albumin data were not available
* patients with incomplete data

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The medical records of 39,135 enrolled trauma patients registered between January 1, 2009 and December 31, 2019 were reviewed for this study (Figure 1). The enrolled patients experienced trauma from different injuries and were hospitalized for treatment. Of the 7,136 patients who were admitted to the ICU, 1,926 older trauma patients were aged ≥ 65 years. After excluding patients whose albumin data were not available and those with incomplete data (n = 1,226), 700 older trauma patients were finally included in the study. Detailed information of the study population was extracted from the Trauma Registry System of the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2020-09-14 (Actual); Study Completion 2020-09-20 (Actual)

PRIMARY OUTCOMES:
Mortality outcome | through study completion, an average of 1 month
  Mortality outcome of older trauma patients in the ICU.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan